CLINICAL TRIAL: NCT06852066
Title: Comparison of Local Anesthetic Techniques on Pain, Anxiety and Hemodynamic Changes in Mandibular Impacted Third Molar Surgery
Brief Title: Comparison of Computer-Assisted and Conventional Local Anesthesia Methods in Mandibular Impacted Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, İsmail Çalışkan, Research Assistant, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ICaliskan96
Record Dates: First submitted 2025-02-07; First posted 2025-02-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-02

CONDITIONS: Molar, Third; Surgery, Oral; Anxiety; Local Anesthesia; Hemodynamic Changes; Comparison of the Efficacy; Computer Assisted Local Anesthesia
Keywords: Ccomputer assisted local anesthesia; Conventional local anesthesia; Wisdom tooth; Surgery; Anxiety; Hemodynamic changes
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 1. Computer-Assisted Local Anesthesia Group (Arm 1)
     Participants in this group will receive computer-assisted local anesthesia using the SleeperOne5 (Dental Hi Tec, Cholet, France) system. The anesthetic used will be 2% articaine with 1:100,000 epinephrine. Injection will be performed under controlled pressure, with an administration duration of 60 seconds.
     Inferior alveolar nerve block and supplemental buccal anesthesia will be applied.
  2. Conventional Local Anesthesia Group (Arm 2)
  Participants in this group will receive conventional local anesthesia using a standard dental syringe (40 mm 27G needle) under manual pressure. The anesthetic used will be 2% articaine with 1:100,000 epinephrine. The injection duration will be 30 seconds under manual pressure. Inferior alveolar nerve block and supplemental buccal anesthesia will be applied.
Who Masked: Participant
Masking Description: There are 2 groups in our study, the first study group will be anesthetized with computer-assisted local anesthesia and the second study group will be anesthetized with conventional local anesthesia. A researcher who is not directly involved in the surgeries or evaluations will perform the randomization procedure. Sequentially numbered envelopes will be used, each containing the technique and the side to be operated on first. Before the local anesthesia injection, the patient's eyes will be closed and the sound of the computer-assisted anesthesia device will be suppressed. These procedures will be performed so that the patients are unaware of the randomly selected technique when local anesthesia is administered, thus ensuring study blindness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Computer-Assisted Local Anesthesia (Experimental): Description: Participants in this arm will receive computer-assisted local anesthesia before undergoing impacted mandibular third molar extraction.
  Interventions Assigned: Computer-Assisted Local Anesthesia
  Interventions: Procedure: Computer-Assisted Local Anesthesia
- Arm 2: Conventional Local Anesthesia (Experimental): Description: Participants in this arm will receive conventional local anesthesia before undergoing impacted mandibular third molar extraction.
  Interventions Assigned: Conventional Local Anesthesia
  Interventions: Procedure: Conventional Local Anesthesia

INTERVENTIONS:
Procedure: Computer-Assisted Local Anesthesia — Description: Local anesthesia applied using the SleeperOne5 (Dental Hi Tec, Cholet, France) device, with controlled injection speed (60 seconds).
  Drug Used: 2% Articaine with 1:100,000 Epinephrine Needle Type: 35 mm, 30G dental syringe
  Arms: Arm 1: Computer-Assisted Local Anesthesia
Procedure: Conventional Local Anesthesia — Description: Local anesthesia applied using a manual dental syringe, with injection speed manually controlled (30 seconds).
  Drug Used: 2% Articaine with 1:100,000 Epinephrine Needle Type: 40 mm, 27G dental syringe
  Arms: Arm 2: Conventional Local Anesthesia

SUMMARY:
The goal of this clinical trial is to evaluate the effects of computer-assisted local anesthesia and conventional local anesthesia on pain perception and dental anxiety during inferior alveolar block anesthesia in impacted mandibular third molar surgeries with bone retention. The study also aims to assess the impact of anesthesia techniques on physiological parameters during the procedure.

The main questions it aims to answer are:

Does computer-assisted local anesthesia reduce pain perception compared to conventional local anesthesia? What are the effects of both anesthesia techniques on dental anxiety and vital signs (systolic/diastolic blood pressure, pulse rate, oxygen saturation, and respiratory rate) during the procedure?

Participants who meet the inclusion criteria will undergo impacted mandibular third molar extractions under two different anesthesia techniques:

One group will receive computer-assisted local anesthesia. The other group will receive conventional local anesthesia. Anxiety and pain measurements will be recorded during the anesthesia administration and throughout the surgical procedure. Vital signs, including systolic and diastolic blood pressure, pulse rate, oxygen saturation, and respiratory rate, will be monitored and compared between the study groups.

This study aims to provide insights into improving pain management and patient comfort during oral surgical procedures.

DETAILED DESCRIPTION:
This clinical trial aims to compare the effects of computer-assisted local anesthesia and conventional local anesthesia on pain perception, dental anxiety, and physiological responses during inferior alveolar nerve block in impacted mandibular third molar surgeries with bone retention. The study evaluates whether the computer-assisted anesthesia technique provides better pain control and reduces anxiety compared to the conventional technique.

Study Design This is a randomized, single-blind clinical trial involving 40 participants who meet the inclusion criteria. Each participant will undergo bilateral, symmetrical impacted mandibular third molar extractions. One side will be anesthetized using computer-assisted local anesthesia, while the other side will receive conventional local anesthesia. A researcher uninvolved in the surgeries will conduct the randomization, using sequentially numbered envelopes to determine the technique and the side to be operated on first. Participants will be blinded to the anesthesia technique used during the procedure.

Anesthesia Protocol Inferior alveolar nerve block and supplemental buccal anesthesia will be applied in both study groups.

Conventional Local Anesthesia: Administered with a 40 mm 27G dental syringe under manual pressure.

Computer-Assisted Local Anesthesia: Performed using the SleeperOne5 (Dental Hi Tec, Cholet, France) system with a 35 mm 30G syringe under controlled pressure.

The anesthetic solution in both groups will be 2% articaine with 1:100,000 epinephrine. The maximum amount administered will be 2 cartridges for the computer-assisted group and 2 ampoules for the conventional group per session. Injection speed is fixed at 60 seconds for the computer-assisted group, while in the conventional group, it will be administered in 30 seconds. The inferior alveolar nerve block will be performed by a single surgeon for all patients to ensure standardization.

Surgical Procedure

A standardized impacted third molar extraction procedure will be performed for all participants. The steps are as follows:

Incision and Flap Elevation: A No. 15 scalpel blade will be used to create an envelope flap incision in the mucosa. The flap will be elevated with a periosteal elevator.

Bone Removal: Access to the impacted tooth will be achieved through bone removal using a surgical micromotor (NsK model, 40,000 rpm) with a steel round or fissure bur under continuous sterile saline irrigation.

Tooth Extraction: Following osteotomy and tooth sectioning (if needed), the impacted tooth will be extracted.

Wound Closure: The flap will be repositioned and sutured using 3/0 atraumatic silk sutures (16 mm, 3/8 round needle).

The surgical protocol will be identical in both groups, ensuring no variability in the procedure itself.

Pain and Anxiety Assessment

Multiple validated scales will be used to assess pain, anxiety, and patient perception of the procedure at different time points:

Before and after anesthesia administration:

Dental Anxiety Scale State-Trait Anxiety Inventory (STAI) Modified Dental Anxiety Scale (MDAS) Amsterdam Preoperative Anxiety Scale (APAIS) Dental Fear Scale (DKS) Visual Analog Scale (VAS)

Immediately after the surgery:

Postoperative versions of the above scales Postoperative satisfaction questionnaire Physiological Measurements

During the study, vital signs will be monitored at predefined time intervals:

Systolic and diastolic blood pressure Pulse rate Oxygen saturation Respiratory rate

These parameters will be recorded at the following time points:

Before anesthesia administration During local anesthesia injection During each step of the surgery (incision, osteotomy, extraction, suturing) After the procedure Postoperative Care

All patients will be prescribed a standard postoperative regimen, including:

Antibiotics (Penicillin or Clindamycin) NSAID pain relievers (Naproxen sodium) Chlorhexidine gluconate mouthwash Instructions for a soft diet and maintaining oral hygiene Statistical Analysis Sample size was determined using G*Power 3.1.9.4 software. Based on an effect size of 0.35, Type I error of 0.05, and statistical power of 80%, the required sample size was calculated as 35 participants. To account for potential exclusions, 40 participants will be included.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in the study:

* Must be between 18 and 40 years old
* Must have bilaterally impacted mandibular third molars with bone retention
* Impacted teeth must be at a mesioangular angle, classified as Class 1-2 and A--B type (Pell & Gregory classification)
* Must have an impacted tooth difficulty level of 3-5 according to the Pederson Difficulty Index
* Must be classified as ASA 1 (healthy individuals with no systemic diseases)
* Must be able to read and understand questionnaire forms and provide informed consent Must voluntarily agree to participate in the study and sign the informed consent form

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

* Presence of any systemic disease (e.g., cardiovascular disease, liver disease, hematologic disorders, neoplastic diseases, rheumatic conditions, diabetes mellitus)
* History of psychiatric disorders or current use of anxiolytics, antidepressants, or anticonvulsants
* Use of anti-inflammatory, analgesic, or anxiolytic medications prior to the procedure that could affect pain, inflammation, or anxiety responses
* Chronic medication use, including antihistamines, NSAIDs, steroids, or antidepressants
* Presence of oral pathologies affecting pain perception (e.g., pulpitis, periodontitis, oral ulcers, cysts, or tumors)
* Suspected or confirmed pregnancy or breastfeeding
* Allergy to the local anesthetic (articaine) used in the study
* Hearing impairment that could interfere with study participation
* Presence of dentophobia (severe dental phobia)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | During surgery, at the following time points: Before local anesthesia injection, Immediately after surgery
  The anxiety levels will also be recorded on a visual analog scale, which has been shown to be a valid way to assess dental anxiety. This scale consists of a 100 mm horizontal line drawn on paper, the left end of which is marked as "no anxiety at all", the right end as "worst anxiety imaginable", and there is no other expression or number on the line. On the other hand, since pain is a condition that varies from person to person, objective measurement is not possible. This scale is used to numerically record the pain intensity that the patient feels at that moment, which cannot be measured numerically. It is also one of the most commonly used methods in the assessment of pain. The patient is asked to mark/express their pain on a 10 cm long line. "0" means no pain, "10" means severe pain. There are levels on the scale from "no pain" to "unbearable pain". It is the most commonly used verbal pain scale.
Modified Dental Anxiety Scale (MDAS) Score | Before local anesthesia injection (Baseline), Immediately after surgery
  Developed by Corah and is the most commonly used scale to measure dental anxiety, the modified version of DAS (MDAS) is preferred more. MDAS consists of a total of 5 questions. When the entire scale is evaluated, the lowest possible score is 5 and the highest is 25. Studies conducted in Turkey have reported that the scale is valid and reliable. The dental anxiety threshold for MDAS is accepted as ≥ 15. Scores of 19 and above indicate severe anxiety. In addition to C-DAS, it includes a question about local anesthetic injection. Since injection is effective on anxiety and phobia, it can be said that MDAS is more advanced.
  Unit of Measure: MDAS Score (5 to 25) Scale Information: Higher scores indicate higher dental anxiety.
Dental Fear Scale (DKS) Score | Before local anesthesia injection (Baseline), Immediately after surgery
  The Dentistry Fear Scale was developed by Kleinknecht et al. in 1973 to examine the level of fear towards various procedures in dentistry. The responses to these questions in this scale, which includes 20 questions aimed at determining the level of fear and tension regarding dental procedures, are scored between 1-5 (Likert type) and a total value between 20-100 is obtained. This scale has 20 items reflecting many symptoms of dental fear and anxiety. Two items focus on avoidance, 5 items focus on physiological arousal, 12 items assess fear towards specific dental stimuli and the last item observes general fear. Scores of 63 and above indicate high anxiety values.
  Unit of Measure: DKS Score (20 to 100) Scale Information: Higher scores indicate greater dental fear.
State-Trait Anxiety Inventory (STAI) Score | Before local anesthesia injection (Baseline), Immediately after surgery
  Spielberger's "State-Trait Anxiety Inventory" (STAI) scale is another scale used in the pre-procedure anxiety assessment. Scores on the 20-question scale range from 1 (not at all) to 4 (completely). Positive scores (increasing the total anxiety score) are given for items 3, 4, 6, 7, 9, 12, 13, 14, 17, and 18 on the scale, and negative scores (decreasing the total anxiety score) are given for items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The highest score is 80, and the lowest score is 20. A high total score is an indication that the person's anxiety level is also high. STAI is a highly reliable, easy-to-implement, and easy-to-evaluate scale that can be used to assess feelings of anxiety, tension, and nervousness momentarily; and anxiety predisposition.
  Unit of Measure: STAI Score (20 to 80) Scale Information: Higher scores indicate higher anxiety levels.
Amsterdam Preoperative Anxiety Scale (APAIS) Score | Before local anesthesia injection (Baseline), Immediately after surgery
  The Amsterdam Preoperative Anxiety and Information Scale (APAIS) was developed by the Moermann group in the Netherlands in 1996. It is one of the tests used to assess preoperative anxiety. The source of anxiety is divided into three in this test: anxiety about surgery, anxiety about anesthesia, or anxiety caused by lack of information. In order to objectify the survey, a numerical value based on a 5-point Likert scale is given to each statement according to severity; 1=none, 2=mild, 3=moderate, 4=severe, 5=extreme severity. Anesthesia anxiety is calculated by adding the scores given to questions 1 and 2, surgical anxiety to questions 4 and 5, and the total anxiety score is calculated by adding both. The statements expressing the desire to learn about anesthesia and surgery are questions 3 and 6. The lowest score is 6, and the highest score is 30.
  Unit of Measure: APAIS Score (6 to 30) Scale Information: Higher scores indicate greater preoperative anxiety.

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure Changes | Before local anesthesia injection (Baseline) Immediately after local anesthesia injection During surgery at key procedural steps (incision, osteotomy, extraction, suturing) Immediately after surgery
  Blood pressure levels (systolic and diastolic) will be measured at predefined time points during the procedure.
  Unit of Measure: mmHg
Pulse Rate Changes | Before local anesthesia injection (Baseline) Immediately after local anesthesia injection During surgery at key procedural steps (incision, osteotomy, extraction, suturing) Immediately after surgery
  Pulse rate will be recorded at multiple stages of the procedure to evaluate autonomic nervous system response.
  Unit of Measure: Beats per minute (bpm)
Oxygen Saturation Levels (SpO₂) During Surgery | Before local anesthesia injection (Baseline) Immediately after local anesthesia injection During surgery at key procedural steps (incision, osteotomy, extraction, suturing) Immediately after surgery
  Oxygen saturation will be monitored throughout the procedure to assess potential stress responses and hypoxia risks.
  Unit of Measure: Percentage (%)
Respiratory Rate Changes | Before local anesthesia injection (Baseline) Immediately after local anesthesia injection During surgery at key procedural steps (incision, osteotomy, extraction, suturing) Immediately after surgery
  Respiratory rate will be recorded at multiple time points to evaluate physiological responses to different anesthesia techniques.
  Unit of Measure: Breaths per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Sciences University, Faculty of Dentistry, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The medical condition investigated in our study is to reduce the pain sensation that occurs during local anesthetic injections in patients who need impacted wisdom tooth surgery and to measure the changes in anxiety, pain levels and vital values of patients during impacted wisdom tooth surgeries. This study aims to comparatively measure the effects of computer-assisted local anesthesia and conventional local anesthesia on dental anxiety and pain during bone retention impacted wisdom tooth surgeries when inferior alveolar block anesthesia is applied, as well as the effects of anesthesia techniques on the depth of the operation during the operation.

REFERENCES:
- [Background] Ozer S, Yaltirik M, Kirli I, Yargic I. A comparative evaluation of pain and anxiety levels in 2 different anesthesia techniques: locoregional anesthesia using conventional syringe versus intraosseous anesthesia using a computer-controlled system (Quicksleeper). Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Nov;114(5 Suppl):S132-9. doi: 10.1016/j.oooo.2011.09.021. Epub 2012 May 6. PMID 23063389
- [Background] Libonati A, Nardi R, Gallusi G, Angotti V, Caruso S, Coniglione F, Marzo G, Mattei A, Tecco S, Paglia L. Pain and anxiety associated with Computer-Controlled Local Anaesthesia: systematic review and meta-analysis of cross-over studies. Eur J Paediatr Dent. 2018 Dec;19(4):324-332. doi: 10.23804/ejpd.2018.19.04.14. PMID 30567452
- [Background] Araujo GM, Barbalho JC, Dias TG, Santos Tde S, Vasconcellos RJ, de Morais HH. Comparative Analysis Between Computed and Conventional Inferior Alveolar Nerve Block Techniques. J Craniofac Surg. 2015 Nov;26(8):e733-6. doi: 10.1097/SCS.0000000000002245. PMID 26594989